CLINICAL TRIAL: NCT03431103
Title: The Effect of Exercise on Systemic Inflammation in Veterans With COPD and OSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Salem Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MM 0013
Record Dates: First submitted 2017-12-21; First posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: COPD; OSA; Home Exercise; Inflammation
Keywords: overlap; exercise; inflammation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Inflammation; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- After home exercise program (Other): Patients will be instructed to use the Wii Fit for 20 minutes at least twice a week for 12 weeks using specific Wii Fit exercises while on the Wii pressure sensor floor mat. The Wii Fit exercises will be as follows: 1." Basic Run" (warm-up exercise by walking in place); 2."Bird's Eye, Bull's-Eye" (mostly arms, requires arm flipping); 3."Free Step" (lower extremity exercise); 4."Hula Hoop" (gyration exercise)
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — 12 week home exercise program

SUMMARY:
The overlap syndrome (OS), i.e. the association of both Chronic Obstructive Pulmonary Disease (COPD) and Obstructive Sleep Apnea (OSA) in a single Veteran, is prevalent and associated with increased cardiovascular disease (CVD) morbidity. Home-based exercise interventions that translate to a lifestyle with increased physical activity (PA) are an ideal strategy as 150 minutes of leisure time PA a week is associated with a significant reduction in risk of CVD related events and death. This novel research study will help develop a home exercise intervention that is largely accepted by OS Veterans, as a first step toward implementing PA into the routine medical care of the large Veteran population with COPD and OSA. This data will be used for larger studies on CVD risk and its modification with exercise in OS, a research area that is urgently needed given its high impact on Veterans' morbidity, mortality and health-care associated costs.

DETAILED DESCRIPTION:
The term "overlap syndrome" (OS) is used to describe the association of both chronic obstructive pulmonary disease (COPD) and obstructive sleep apnea disease (OSA) in a single Veteran. Given the high prevalence of both COPD and OSA, it is expected that a third of Veterans with OSA could be affected by OS. Importantly, Veterans with OS have a higher cardiovascular morbidity and mortality than either OSA or COPD-only Veterans, likely due to worse nocturnal hypoxia and subsequent inflammation and endothelial dysfunction. Therefore, therapy for Veterans with OS that decreases cardiovascular disease (CVD) by targeting inflammation is a high priority. Home-based exercise interventions that translate to a lifestyle with increased physical activity (PA) are an ideal strategy as 150 minutes of leisure time PA a week is associated with reduction in risk of CVD-related events and death. Further, PA decreases biomarkers of systemic inflammation. However, no data is available on the effect of exercise on biomarkers of systemic inflammation in Veterans with OS. It is difficult to increase the leisure time PA in adults with COPD and OSA as this population is more sedentary due to a combination of increased obesity, daytime sleepiness and dyspnea. Therefore, home-based exercise would be ideal for these Veterans. The objective of this proposal is to conduct a single arm 12-week home-based exercise pilot intervention to determine the effect on biomarkers of systemic inflammation in 50 Veterans with OS on CPAP. The investigator hypothesizes that 1) Baseline PA intensity and duration will correlate inversely with the biomarkers of systemic inflammation independently of nocturnal hypoxia; and 2) Exercise training using a home-based computer exercise program will decrease biomarkers of systemic inflammation and increase exercise capacity in Veterans.

ELIGIBILITY:
Inclusion Criteria:

* Veterans from the Salem VAMC pulmonary clinics will be screened for a diagnosis of OSA and treatment with CPAP therapy. In addition, an inclusion criterion also will be a recent PFT diagnostic of COPD (FEV1/FVC <0.7 and FEV1< 80%). Only Veterans with OS who are compliant with CPAP therapy will be enrolled in the study.

Exclusion Criteria:

* orthopedic problems, fall-risk, balance problems;
* any regular participation in structured exercise sessions;
* other concomitant sleep disorder;
* unstable cardiovascular or pulmonary disease;
* acute infectious illness in the prior month;
* hospitalization in prior month;
* prescription of systemic glucocorticoids or immune-suppressive agents in the prior month and
* weight above 330 pounds, the limit allowed by the Wii pressure sensor floor mat.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-12-05 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
To assess the relationship between baseline physical activity (meters obtained from 6 minute walk test) and serum hs-CRP (mg/L) | 24 months
  We will measure baseline physical activity (meters obtained from 6 minute walk test) and serum hs-CRP (mg/L) prior to the home-based computer exercise program (Wii Fit)

SECONDARY OUTCOMES:
To determine the impact of a 12-week home-based Wii Fit exercise program on physical activity (meters obtained from 6 minute walk test) and serum hs-CRP (mg/L) | 3 months
  Physical activity (meters obtained from 6 minute walk test) and serum hs-CRP (mg/L) will be measured before and after a 12-week home-based Wii Fit exercise program

CONTACTS AND LOCATIONS:
Locations (1):
- Salem VAMC, Salem, Virginia, United States

IPD SHARING:
Plan to Share IPD: No